CLINICAL TRIAL: NCT03176589
Title: Effect of PEP on Oxygen Saturation and Carbon Dioxide After Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Karl A Franklin, Ass Prof, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/195-31
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Blood Gas Monitoring, Transcutaneous
Keywords: positive expiratory pressure; oxygen saturation; abdominal surgery; carbon dioxide
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: Positive expiratory pressure (PEP) therapy
Who Masked: Care Provider, Outcomes Assessor
Masking Description: tube without resistance is given to patients. Randomization order is given after the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sham PEP (Sham Comparator): 3 cycles of 10 deep inspiration and expiration in a sham tube without expiratory resistance
  Interventions: Device: Placebo comparator, Deep inspiration and expression in a placebo tube without resistance
- PEP (Active Comparator): 3 cycles of 10 deep inspiration followed by expiration with positive expiratory pressure (PEP) device or PEP bottle of 10-15 cm of water pressure
  Interventions: Device: positive expiratory pressure (PEP)
- deep breathing maneuvers (Experimental): 3 cycled of 10 deep breathing maneuvers without PEP or sham PEP
  Interventions: Other: Deep breathing maneuvers

INTERVENTIONS:
Device: positive expiratory pressure (PEP) — Patients take a deep inspiration followed by PEP expiration with an expiratory pressure of 10-15 cm H2O
  Arms: PEP
Device: Placebo comparator, Deep inspiration and expression in a placebo tube without resistance — Deep inspirations 3 times 10 and expiration in a placebo tube without expiratory resistance
  Arms: sham PEP
Other: Deep breathing maneuvers — deep breathing maneuvers 3 times 10 breahs without any device at expiration
  Arms: deep breathing maneuvers

SUMMARY:
Positive expiratory pressure( PEP) is routinely given to patients after surgery in order to improve lung function and oxygen saturation. There is, however, no evidence of effect on lung function, postoperative pneumonia or any other outcome (Guimarães MMF, Tyson AF). The investigators aim to test the immediate effects of PEP therapy on oxygen saturation and carbon dioxide after abdominal surgery. 80 patients will be investigated in RCT design with expiration using PEP or with expiration to a sham-PEP, a tube without resistance. At the end of the study we will also measure the effect of 10x3 deep breathing maneuvers without PEP or shamPEP. Primary outcome: Maximum and minimum levels of continuously measured oxygen saturation from pulse oximetry and transcutaneous carbon dioxide partial pressure during the trial.

DETAILED DESCRIPTION:
Background Hypoxia, reduced lung function and atelectais are common after abdominal surgery and can be hazardous in patients with chronic hypoxia. Positive expiratory pressure (PEP) therapy or incentive spirometry are routinely given to patients after abdominal surgery to counteract atelectasis and improve oxygen saturation. Patients are instructed by a physiotherapist to take deep inspiratory breaths and expire in a PEP-device or PEP bottle. The method is used routinely in Swedish hospital and the patient breathes against 10-15 cm water resistance. This is repeated 10x3 ie 10 deep breaths and exhalation towards PEP then rest, breath, rest and another 10 breaths. This procedure should be done once an hour after surgery. The idea is that this will widen alveoli and abolish atelectasis, thus increasing the oxygen uptake and reducing the risk of postoperative complications.

There is no evidence of effect of PEP and incentive spirometry on postoperative pulmonary complications after abdominal surgery (Guimarães MMF, Tyson AF). Nevertheless, PEP therapy is used in Sweden and internationally. There were no studies found reporting the immediate effect of PEP on continuous oxygen saturation and carbon dioxide partial pressure after surgery.

Aims

What effect does PEP have on oxygen saturation and carbon dioxide partial pressure? What is the effect of deep breathing maneuvers on oxygen saturation and carbon dioxide partial pressure?

Methods

Inclusion: 80 adult patients over 18 years of age who have undergone open or laparoscopic abdominal surgery. Patients receiving postoperative PEP are asked to participate in the study at one or two days after after abdominal surgery.

Exclusion: Patients who cannot participate in using PEP or who do not agree to participate in the study.

Power calculation:.It was estimated that 34 patients were needed to detect a mean (SD) difference in oxygen saturation of 1% (2%) and to detect a difference in transcutaneous PCO2 of 0.5 kPa (1 kPa) with a significance of p < 0.05 and a power of 80%.

Design / Randomization: RCT study with cross-over design. Patients are randomized using computer programs, handled by a person outside the study, to either start with either PEP breathing 10x3 or sham-PEP breathing 10x3.

Method: Starting with lung function assessment to determine PEF (Mini Wright Clement Clarke). Then, application of continuous transcutaneous PCO2 / SaO2 (SenTec Digital Monitoring System, ResMed) and a respiratory belt around the chest detecting the respiratory rate. Data is recorded with computer equipment (Noxturnal T3, ResMed).

The patients are randomized to initiate with either 10x3 breaths using PEP therapy or 10x3 breaths using Sham PEP. After a rest period, patients switch to the second treatment (cross-over). At the end of the trial, all patients take 10X3 deep breaths without PEP or sham PEP.

At the start of the study, baseline level for SaO2 and TcPCO2 is recorded, and an arterial blood gas is recorded to calibrate the transcutaneous PCO2 measurement. Thereafter, the registration continues during breathing / blowing until the patient returns to its baseline values. New PEF examination is made after each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who have undergone open or laparoscopic abdominal surgery.
* Patients receiving postoperative PEP are asked the day after surgery if they want to participate in the study.

Exclusion Criteria:

* Patients who cannot participate in using PEP or who do not agree to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Transcutaneous blood gas measurements: transcutaneous pCO2 | once, within one hour
  transcutaneous pCO2

SECONDARY OUTCOMES:
Pulse oximetry: oxygen saturation (SaO2) | once, within one hour
  oxygen saturation (SaO2)
Lung function: PEF | once, within one hour
  Peak expiratory flow

CONTACTS AND LOCATIONS:
Overall Officials: Karl Franklin, Ass Prof, Principal Investigator — Umea University
Locations (1):
- Dept of Surgery, Inst of Surgical and Perioperative sciences, Umeå, Umea, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guimaraes MM, El Dib R, Smith AF, Matos D. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006058. doi: 10.1002/14651858.CD006058.pub2. PMID 19588380
- [Background] Tyson AF, Kendig CE, Mabedi C, Cairns BA, Charles AG. The effect of incentive spirometry on postoperative pulmonary function following laparotomy: a randomized clinical trial. JAMA Surg. 2015 Mar 1;150(3):229-36. doi: 10.1001/jamasurg.2014.1846. PMID 25607594